

Craven House, West Street, Farnham, Surrey, GU9 7EN

IRAS ID: 234710

Study Site (address and Telephone): \_\_\_\_\_\_

Study Number: TRTN-501

Participant Identification Number for this study: \_\_\_\_\_\_

## **INFORMED CONSENT FORM**

**STUDY TITLE:** An evaluation of The Fitting Success Rate of Senofilcon A soft Contact Lenses in Three Designs

| PARTICIPANT'S STATEMENT | |
|---|---|
| 1. | I confirm that I have read the information sheet dated 17 <sup>th</sup> November 2017 (version 3) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason and without my future care or legal rights being affected. |
| 3 | I agree that anonymised photographs and/or videos may be taken of my eyes, if needed. I understand that these may be necessary to document my ocular health and, aside from my right to withdraw consent from the study entirely, are not optional. |
| 4. | I understand and give permission for my ophthalmic records (eye clinic notes) and research data to be looked at by responsible individuals from the sponsor company, Visioncare Research or from regulatory authorities where it is relevant to my taking part in this research. |
| 5. | I agree to the sponsor company or Visioncare Research Ltd processing my personal data, which I have supplied, and I understand that my anonymised data will be used to support other research in the future and may be shared anonymously with other researchers I further agree to the sponsor company or Visioncare Research Ltd processing personal data about me described as sensitive data within the meaning of the Data Protection Act 1998. |
| 6. | I understand that I am able to obtain a summarised copy of the final study results if I wish and can obtain these by contacting the investigator at the end of the study. |
| 7. | I voluntarily agree to take part in this study and I will get a signed copy of this form, and the information sheet, for my records. |

## VISIONCARE RESEARCH LTD



Craven House, West Street, Farnham, Surrey, GU9 7EN

| Printed Name of Participant | |
|---|---|
| Signature of Participant / Date | .1 |
| attest that the participant had enough time to consicquestions, and voluntarily agreed to be in this study. | ler this information, had an opportunity to ask |
| Printed Name of Person Obtaining Consent | |
| Signature of Person Obtaining Consent / Date | ./ |
| Printed Name of Principal Investigator or Sub-Investiga o waive, if the person obtaining consent is the Principal Investigator or Sub-Investigator or Sub-Investigat | |
| | _ /<br>Date |
| <ul><li>waive, if the person obtaining consent is the Principle</li></ul> | |

TRTN-501 ICF v2 06.Nov.2017